CLINICAL TRIAL: NCT02494375
Title: Sleep and Glycemic Control in Type 1 Diabetic Children
Brief Title: Sleep and Type 1 Diabetes
Acronym: SLEEPT1D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL15_0219
Record Dates: First submitted 2015-07-03; First posted 2015-07-10 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Type 1 Diabetes
Keywords: Sleep; glycemic control; type 1 diabetes; amylase; body composition; lean; overweight; obese
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Overweight; Obesity | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleep and glucose assessement. (Experimental)
  Interventions: Other: Sleep and glucose assessments

INTERVENTIONS:
Other: Sleep and glucose assessments — Sleep characteristics, glycemic control, salivary amylase and body composition will be assessed 3 times, at 3-4 months intervals

SUMMARY:
The primary goal of the study is to determine whether insufficient sleep is associated with poor glycemic control in type 1 diabetic children. Secondary goals aim to determine whether salivary amylase could be an easily accessible and non-invasive biomarker of sleep loss and somnolence, and whether insufficient sleep is linked to body composition. Sleep characteristics, glycemic control, salivary amylase and body composition will be assessed 3 times, at 3-4 months intervals, in 82 type 1 diabetic children.

ELIGIBILITY:
Inclusion Criteria:

- Female and male type 1 diabetic children and adolescents who are followed at the Woman, Mother and Child's Hospital (Hôpital Femme Mère Enfant : HFME) of Bron, France.

Exclusion Criteria:

* Refusal of consent of the parents or the child or the adolescent
* Pregnancy
* Concomitant pathology that severly impacts sleep
* Implanted electrical stimulation device
* Diagnosis of type 1 diabetes <1 year

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2015-06-28 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Association between HbA1c and sleep characteristics | Month 3, Month 6 and Month 9

SECONDARY OUTCOMES:
Glucose levels | Month 3, Month 6 and Month 9
  3 daily pre- and post- meal glucose levels over a 3-day period
Daily salivary amylase variation (Enzyme Activity) | Month 3, Month 6 and Month 9
  Assessment of salivary amylase levels
Body composition (BMI fat and lean mass percentage) | Month 3, Month 6 and Month 9
  Assessment of body composition

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France